CLINICAL TRIAL: NCT00685932
Title: Mobius Pain Study: A Randomized Controlled Trial of Standard Versus Mobius® Retraction at Cesarean Delivery
Brief Title: Mobius® Post-cesarean Pain Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbey Hardy-Fairbanks (Other)
Collaborators: Apple Medical Corporation (Industry)
Responsible Party: Sponsor-Investigator, Abbey Hardy-Fairbanks, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21107
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Results first posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Complications; Cesarean Section; Pregnancy
Keywords: Postpartum pain; Post-cesarean pain; Surgical retractor; Elastic retractor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): This arm will be randomly assigned to have conventional retractions (ie Rich retractors and similar) used in the usual fashion during the cesarean procedure.
- Mobius (Experimental): This arm will be randomized to have the providers who are performing the cesarean section use the Mobius retractor during the cesarean section procedure after the peritoneal cavity is opened.
  Interventions: Device: Mobius Retractor

INTERVENTIONS:
Device: Mobius Retractor — The Mobius retractor is a dual ring elastic self retaining retractor that is inserted into the abdominal cavity after the peritoneal incision has been established. It is then left in place during the hysterotomy incision, delivery of the fetus, hysterotomy repair, inspection and irrigation.
  Arms: Mobius

SUMMARY:
The purpose of this study is to investigate whether the use of the Mobius® retractor decreased post-operative pain after cesarean section verses conventional retractor use. Based on clinical experience and a pilot study, we suspect that the retractor will decrease overall pain as well as lateral pain.

DETAILED DESCRIPTION:
This is a prospective, randomized, patient blinded trial of standard surgical retraction versus Mobius® retraction at cesarean delivery. Women will be approached by their provider at their 36 week prenatal visit regarding potential study participation. They will be given a letter describing the study. If a woman is interested, she will be contacted by a study nurse who will obtain informed consent. Ideally, women will be approached prior to the onset of labor or date of scheduled cesarean delivery so as to provide adequate time to review the study and ask questions. Women who undergo antenatal admission will be also approached by their provider regarding possible study participation and given a recruitment letter. If they are interested, then a study nurse will obtain informed consent.

Consenting women will be randomized after the decision to deliver by cesarean section is made. Randomization will be performed in blocks to control for scheduled versus unscheduled cesarean deliveries using a random numbers generator. Assignments will be kept in sequentially number opaque envelopes. Women will not be informed of their assignment until after discharge from the hospital. Efforts will be made in the operating room to avoid disclosing group assignment and the consent forms will not contain the specific name of the retractor under study. The operative team will be aware of group assignment.

Participants will complete a 7 item pain scale each post-operative day until discharge. This pain scale has been used in a pilot study and found to be accurate. The pain scale is a single page and takes less than 5 minutes to complete.

Charts will be reviewed to obtain clinical information which may have an impact on post-operative pain. This includes information about current and past substance abuse. Because of the increased amounts of post-operative pain experienced by women who use methadone during pregnancy, this group of women will be excluded from the study. To protect the information regarding substance abuse, a certificate of confidentiality has been obtained from the NIH.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Potential for having a cesarean section (scheduled or unscheduled) at Dartmouth Hitchcock Medical Center

Exclusion Criteria:

* Less than 18 years old
* Unable to consent due to language barrier or psychiatric illness
* Current methadone use for chronic pain
* Stat cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Lauria, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Background] Rafique Z, Shibli KU, Russell IF, Lindow SW. A randomised controlled trial of the closure or non-closure of peritoneum at caesarean section: effect on post-operative pain. BJOG. 2002 Jun;109(6):694-8. doi: 10.1111/j.1471-0528.2002.00153.x. PMID 12118650
- [Background] Chanrachakul B, Hamontri S, Herabutya Y. A randomized comparison of postcesarean pain between closure and nonclosure of peritoneum. Eur J Obstet Gynecol Reprod Biol. 2002 Feb 10;101(1):31-5. doi: 10.1016/s0301-2115(01)00503-6. PMID 11803097
- [Background] Giacalone PL, Daures JP, Vignal J, Herisson C, Hedon B, Laffargue F. Pfannenstiel versus Maylard incision for cesarean delivery: A randomized controlled trial. Obstet Gynecol. 2002 May;99(5 Pt 1):745-50. doi: 10.1016/s0029-7844(02)01957-9. PMID 11978282
- [Background] Kadir RA, Khan A, Wilcock F, Chapman L. Is inferior dissection of the rectus sheath necessary during Pfannenstiel incision for lower segment Caesarean section? A randomised controlled trial. Eur J Obstet Gynecol Reprod Biol. 2006 Sep-Oct;128(1-2):262-6. doi: 10.1016/j.ejogrb.2006.02.018. Epub 2006 Apr 18. PMID 16621227
- [Background] Nafisi S. Influence of uterine exteriorization versus in situ repair on post-Cesarean maternal pain: a randomized trial. Int J Obstet Anesth. 2007 Apr;16(2):135-8. doi: 10.1016/j.ijoa.2006.10.009. Epub 2007 Feb 5. PMID 17276669
- [Background] Dunn EA, O'Herlihy C. Comparison of maternal satisfaction following vaginal delivery after caesarean section and caesarean section after previous vaginal delivery. Eur J Obstet Gynecol Reprod Biol. 2005 Jul 1;121(1):56-60. doi: 10.1016/j.ejogrb.2004.11.010. PMID 15950369
- [Background] Granot M, Lowenstein L, Yarnitsky D, Tamir A, Zimmer EZ. Postcesarean section pain prediction by preoperative experimental pain assessment. Anesthesiology. 2003 Jun;98(6):1422-6. doi: 10.1097/00000542-200306000-00018. PMID 12766652
- [Background] Pan PH, Coghill R, Houle TT, Seid MH, Lindel WM, Parker RL, Washburn SA, Harris L, Eisenach JC. Multifactorial preoperative predictors for postcesarean section pain and analgesic requirement. Anesthesiology. 2006 Mar;104(3):417-25. doi: 10.1097/00000542-200603000-00007. PMID 16508387
- [Background] Thompson JF, Roberts CL, Currie M, Ellwood DA. Prevalence and persistence of health problems after childbirth: associations with parity and method of birth. Birth. 2002 Jun;29(2):83-94. doi: 10.1046/j.1523-536x.2002.00167.x. PMID 12051189
- [Background] Dodd J, Pearce E, Crowther C. Women's experiences and preferences following Caesarean birth. Aust N Z J Obstet Gynaecol. 2004 Dec;44(6):521-4. doi: 10.1111/j.1479-828X.2004.00300.x. PMID 15598289
- [Background] McCarthy M Jr, Chang CH, Pickard AS, Giobbie-Hurder A, Price DD, Jonasson O, Gibbs J, Fitzgibbons R, Neumayer L. Visual analog scales for assessing surgical pain. J Am Coll Surg. 2005 Aug;201(2):245-52. doi: 10.1016/j.jamcollsurg.2005.03.034. PMID 16038823
- See also: Description of Mobius retractor from the manufacturer — https://www.coopersurgical.com/Products/Detail/ob-mobius-self-retaining-c-section-retractor
- See also: Dartmouth-Hitchcock Medical Center home page — http://www.dhmc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: July 2008 to March 2010
Groups:
- Control: Conventional retractions (ie Rich retractors and similar) used in the usual fashion during the cesarean procedure.
- Mobius: Subjects underwent cesarean delivery and the Mobius self-retaining retractor was used as the primary method of retraction during hysterotomy, delivery of infant, hysterotomy repair as well as inspection and irrigation. Other conventional retraction was used for the remainder of the procedure as needed. Decision to abandon use of the Mobius was at the discretion of the primary surgeon.
Period: Overall Study
Arm/Group | Control | Mobius
Started | 76 | 78
Completed | 55 | 58
Not Completed | 21 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Mobius | Total
Number analyzed (Participants) | 76 | 78 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 78 | 154
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (5.7) | 30.3 (5.3) | 30.7 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 78 | 154
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 78 | 154

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants Who Report Asymmetrical Pain on Second Post-operative Day After Cesarean Delivery
Description: Visual analog scale will be used to assess pain on the right or left side of the body with activity.VAS will use a 0-7.5cm range on the right and 0-7.5cm range on the left. This scale is with 0 (or central mark) as no pain and increasing as the subject marks away from the central mark.
Time Frame: 2 days post-operation
Measure: Number; unit: participants
Arm/Group | Control | Mobius
Number analyzed (Participants) | 76 | 78
participants | 33 | 32

2. Primary Outcome: The Degree of Pain With Activity on Post-operative Day Number Two
Description: Visual analog scale (VAS) of pain with activity on a scale of 0-15cm with 0cm: No pain to 15cm: Severe pain.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Mobius
Number analyzed (Participants) | 76 | 78
cm | 6.4 (3.0) | 6.3 (2.9)

ADVERSE EVENTS:
Arm/Group | Control | Mobius
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/78
Other Adverse Events (participants affected / at risk) | 0/76 | 0/78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No